CLINICAL TRIAL: NCT00869596
Title: A Randomized Clinical Trial to Assess the Effects of Inhaled Fluticasone on Sputum Neutrophils After Low-dose Inhaled Endotoxin Challenge in Healthy Subjects
Brief Title: Study of Biomarkers of Airway Inflammation (0000-128)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 0000-128; 2009_565
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Airway Inflammation
Keywords: Sputum inflammatory biomarkers
MeSH Terms: interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: Placebo to fluticasone; Drug: Comparator: Lipopolysaccharide (LPS); Drug: Comparator: albuterol
- 2 (Active Comparator): Fluticasone 440 mcg
  Interventions: Drug: fluticasone propionate; Drug: Comparator: Lipopolysaccharide (LPS); Drug: Comparator: albuterol
- 3 (Active Comparator): Fluticasone 1980 mcg
  Interventions: Drug: fluticasone propionate; Drug: Comparator: Lipopolysaccharide (LPS); Drug: Comparator: albuterol

INTERVENTIONS:
Drug: fluticasone propionate — Single dose of fluticasone 440 mcg (2 x 220 mcg) or 1980 mcg (9 x 220 mcg) by metered dose inhaler in two of three treatment periods
  Arms: 2; 3
Drug: Comparator: Placebo to fluticasone — Single dose of placebo to fluticasone (9 x 0 mcg) by metered dose inhaler in one of three treatment periods
  Arms: 1
Drug: Comparator: Lipopolysaccharide (LPS) — 20,000 EU LPS by inhalation 1 hour postdose of fluticasone or placebo in each of three treatment periods
Drug: Comparator: albuterol — Albuterol two 100 mcg inhalations by metered dose inhaler prior to sputum induction at screening, twice during each of the three treatment periods, and at the post-study follow up visit.

SUMMARY:
This study will evaluate the effects of inhaled fluticasone on cell counts and inflammatory mediators measured in sputum of healthy volunteers following exposure to inhaled lipopolysaccharide.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects who can have children must have a negative pregnancy test at screening and agree to use two methods of birth control throughout the study
* Male subjects with female partner(s) who can have children agree to use an acceptable method of birth control throughout the study
* Subject is a nonsmoker
* Subject is in generally good health
* Subject is willing to comply with the diet, alcohol, and caffeine study restrictions

Exclusion Criteria:

* Subject is a nursing mother
* Subject has taken oral corticosteroids within 8 weeks or inhaled/nasal corticosteroids within 4 weeks of screening
* Subject has nasal polyps, recent nasal surgery, or an ongoing upper or lower respiratory tract infection
* Subject has a recent history of allergic rhinitis at screening
* Subject has any respiratory disease at screening
* Subject has daily phlegm or a chronic cough
* Subject is unable to refrain from the use of any prescription or non-prescription drugs or herbal remedies during the study
* Subject consumes excessive amounts of alcohol or caffeine
* Subject has had major surgery, or donated or lost 1 unit of blood within 4 weeks of screening
* Subject has a history of stroke, seizures, or major neurological disorders
* Subject regularly uses illicit drugs or has a history of drug/alcohol abuse
* Subject received a vaccination within 3 weeks of screening

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2009-03; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Sputum percent neutrophils | 6 hours following inhaled LPS challenge

SECONDARY OUTCOMES:
Sputum absolute neutrophils (per mL) | 6 hours following inhaled LPS challenge
Sputum levels of IL1beta and IL8 | 6 hours following inhaled LPS challenge
Sputum mRNA expression levels of CD14 and IL1beta | 6 hours following inhaled LPS challenge

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC